CLINICAL TRIAL: NCT04204369
Title: Usefulness of a Musculoskeletal Ultrasound Course in an Orthopedic Surgery Residency Training Program
Brief Title: A Musculoskeletal Ultrasound Course for Orthopedic Surgery Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H2017:227 (HS20921)
Record Dates: First submitted 2019-12-15; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Tendon Disorder
Keywords: point of care ultrasound; musculoskeletal ultrasound; sonography; resident education; orthopaedic surgery; online curriculum
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: One group receiving intervention. Assessement prior to intervention, immediately after, and at 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teaching arm (Experimental): This group received the teaching intervention and was evaluated before and after the intervention. Improvement was compared to their performance prior to the intervention.
  Interventions: Other: Ultrasound education curriculum

INTERVENTIONS:
Other: Ultrasound education curriculum — Participants were enrolled in a musculoskeletal ultrasound course including 2 components:
  * An online course (1-2 hours) to be done before the practical session. The videos were made available one (1) month prior to the practical course. This component reviewed the basics of ultrasonography, as well as the normal and abnormal appearance of relevant musculoskeletal structures (bone, tendon, ligaments, muscles, bursas, and nerves), and the ultrasound anatomy of high yield regions of the musculoskeletal system (shoulder, elbow, knee, ankle)
  * A practical session (4-6 hours) done during one of the usual academic days of the orthopedic residency program. This session covered the use of the ultrasound; the examination of the shoulder, elbow, knee, and ankle; ultrasound-guided musculoskeletal injections and aspirations; and ultrasound-guided distal radius fracture reductions. Ample practice time was given to the residents using means such as phantom models, cadavers, and real patients.

SUMMARY:
A group of orthopedic surgery residents underwent a structured online and practical musculoskeletal ultrasound course. Their proficiency on a written and practical exam, as well as frequency and comfort when using was recorded prior to the course, immediately after, and 6 months after the course.

DETAILED DESCRIPTION:
Musculoskeletal ultrasound (MSK-US) can have many uses for orthopedic surgeons, such as assisting in clinical diagnosis for muscle, tendon and ligament injuries, providing direct guidance for joint injections, or assessing the adequacy of a reduction in the emergency department. However, proficiency in sonography is not a requirement for certification in orthopedic surgery in Canada, and orthopedic trainees are rarely exposed to the subject. This project aims assess the usefulness in clinical education of a newly implemented MSK-US course in an orthopedic surgery program.

An MSK-US course for orthopedic surgery residents has been developed. An online survey covering the level of training of the resident, their prior experience with ultrasound (number of times used by month) and their comfort level with different parts of the examination (numeric analog scale - NAS), was filled by the participants prior to the course. A pre-course written and practical test was also given to the residents. Following the course, the participants were reassessed with the same tests and surveys on the same day as the course, and at 6 months post. Change in frequency of use, comfort level and test scores were assessed using a Kruskal-Wallis ANOVA and post-hoc Wilcoxon tests.

It was expected that residents' frequency of use, comfort level and tests scores would improve following the implementation of the course. The results were expected to be maintained at the 6 months endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Be an orthopedic surgery resident
* Training at the University of Manitoba
* Post-graduate year (PGY) one to five

Exclusion Criteria:

* Residents having less than six months of training left before graduation
* Residents on extended leave (for example: completing graduate studies abroad, parental leave, and sabbatical)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Change in Musculoskeletal ultrasound knowledge after the course | Before the course (within a month), immediately after the course (same day)
  A 13 questions written examination was given to the residents using an online platform at each endpoint. The exam covered the basics of ultrasound physics; how to use the machine; the normal and pathologic appearance of tendons, ligaments, and muscles; and ultrasound appearance of the musculoskeletal anatomy described in the course. The score was reported on a scale from 0 to 100, with 100 being the best score.
Change in Musculoskeletal ultrasound knowledge at 6 months | Before the course (within a month), 6 months after the course
  A 13 questions written examination was given to the residents using an online platform at each endpoint. The exam covered the basics of ultrasound physics; how to use the machine; the normal and pathologic appearance of tendons, ligaments, and muscles; and ultrasound appearance of the musculoskeletal anatomy described in the course. The score was reported on a scale from 0 to 100, with 100 being the best score.

SECONDARY OUTCOMES:
Practical shoulder ultrasound exam | Immediately after the course (same day), 6 months after the course
  Each participant underwent a practical examination assessing ultrasound proficiency at each endpoint. The residents were assessed by one of the author of the study on their ability to perform a shoulder ultrasound exam as well as the different tasks related to the MSK-US. For each task, the assessor rated the participant on a scale of 0 to 2, where :
  * 0 means an inability to perform the task,
  * 1 means the task is only partially completed,
  * 2 means that the task that is performed correctly.
  The final score was then be calculated and reported in percentage (with 100 being a perfect score) for the analysis.
Ultrasound comfort in clinical setting | Before the course (within a month), 6 months after the course
  A questionnaire covering different aspect of ultrasound use by the residents was given using the online platform at each endpoint. The questionnaire inquired about the comfort level when using MSK-US for different examinations and procedure (Numeric Analog Scale from 0 to 10, with 0 being very uncomfortable and 10 being very comfortable). Each numeric analog scale was reported independently and not compound score was created:
  * Setting up the ultrasound machine
  * Choosing the appropriate probe
  * Adjusting the depth and contrast
  * Diagnosing a ligament, tendon, muscle, nerve, or bone injury
  * Performing a joint injection or aspiration
  * Performing an injection or aspiration in any other region than a joint
  * Guiding the reduction of a fracture in the forearm
  * Guiding the reduction of any other fracture than the forearm
  * Performing ultrasound in general
Ultrasound use in clinical setting | Before the course (within a month), 6 months after the course
  The questionnaire inquired about the number of time ultrasound was used in the last 6 months for different examinations and procedures. This was reported as an absolute number for each aspect of ultrasound use:
  * Diagnosing a ligament, tendon, muscle, nerve, or bone injury
  * Performing a joint injection or aspiration
  * Performing an injection or aspiration of any other region than a joint
  * Guiding the reduction of a fracture in the adult patient
  * Guiding the reduction of a pediatric fracture

OTHER OUTCOMES:
Socio-demographic questionnaire | Before the course (within a month)
  This questionnaire was presented to participants once at the moment of their inclusion in the study. It covered the residents' level of training (post-graduate year), age, sex, the amount of prior exposure to ultrasound (in approximate hours), and the different settings in which the residents have been exposed to MSK-US.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Larrivee, MD-MSc, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to other researcher. Because of the small size of the orthopedic surgery program, sharing IPD would make identification of individuals unavoidable.